CLINICAL TRIAL: NCT01490554
Title: Effectiveness of Autologous Fibroblast Grafts in the Regeneration of Facial Ectoderm
Brief Title: Autologous Fibroblast Grafts in Facial Skin Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, LYDIA MASAKO FERREIRA, Full Professor and Chairwoman and Head of the Division of Plastic Surgery and Department of Surgery, Federal University of Sao Paulo-UNIFESP, SP, Brazil, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP UNIFESP-1787/07
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Skin Aging
Keywords: Skin aging; fibroblasts; transplantation; autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous fibroblast grafts (Experimental): autologous fibroblast grafts
  Interventions: Procedure: autologous fibroblasts grafts

INTERVENTIONS:
Procedure: autologous fibroblasts grafts — Autologous cultured fibroblasts will be grafted in facial skin

SUMMARY:
The purpose of this study is to evaluate the presence of skin changes after grafting of autologous fibroblasts by means of biophysical, histological, immunohistological, gene expression, glycosaminoglycan, and sensitivity analyses.

DETAILED DESCRIPTION:
- Analytical prospective autocontrolled study

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 50 to 70 years with facial wrinkles (rhytides),
* Fitzpatrick III skin type, and
* Who had reached menopause at least 3 years before entering the study were eligible for participation.

Exclusion Criteria:

* Women with uncontrolled comorbid conditions,
* Smokers,
* Alcohol and corticosteroid users,
* Who had undergone chemical peeling or skin filling in the face or neck at least 12 months prior to the study,
* Who had a keloid scar,
* Who scored below 18 on the Mini-Mental State Examination,
* Who had any psychiatric disorder or those undergoing orthodontic treatment were excluded from the study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Regeneration of facial ectoderm | one year after the grafting of autologous fibroblasts.
  To evaluate the presence of skin changes after grafting of autologous fibroblasts by means of biophysical, histological, immunohistological, gene expression, glycosaminoglycan, and sensitivity analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Ferreira, MD, PhD, Principal Investigator — Federal University of São Paulo